CLINICAL TRIAL: NCT05506215
Title: A Prospective, Multicenter, Open Label, Randomized, Controlled Clinical Study Evaluating the Effect of NovoSorb ® SynPath™ Dermal Matrix Compared to Standard of Care (SOC) In the Treatment of Nonresponsive, Chronic Diabetic Foot Ulcers.
Brief Title: Randomized Clinical Study Comparing SynPath to Standard of Care in Treatment of Chronic Diabetic Foot Ulcers
Acronym: DFUs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After review of study data, sponsor determined wound bed preparation prior to product application was not being followed. A new study will be considered with clearer definition of wound bed preparation and strict adherence to the steps for use.
Sponsor: PolyNovo Biomaterials Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-005
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Foot; Chronic Foot Ulcer; Wound Healing; Foot Ulcer
Keywords: Ulcer; Diabetic; Acellular Dermal Matrix Template; Diabetes Complications
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Ulcer; Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NovoSorb SynPath (Experimental): Arm receives application on NovoSorb SynPath Dermal Matrix and appropriate Off-loading
  Interventions: Device: SynPath Acellular Dermal Matrix plus Off-loading Device
- Standard of Care (Active Comparator): Arm receives application of wound dressing composed of 90% Collagen and 10% Alginate plus appropriate Off-loading
  Interventions: Device: Wound Dressing composed of 90% collagen and 10% Alginate plus Off-loading Device

INTERVENTIONS:
Device: SynPath Acellular Dermal Matrix plus Off-loading Device — Application of SynPath
  Arms: NovoSorb SynPath
Device: Wound Dressing composed of 90% collagen and 10% Alginate plus Off-loading Device — Application Wound Dressing composed of Collagen and Alginate
  Arms: Standard of Care

SUMMARY:
The study will evaluate the efficacy of SynPath™, a synthetic dermal matrix, in the treatment of diabetic foot ulcers in subjects with diabetes mellitus versus Standard of Care treatment.

Half the subjects with be treated using SynPath™ while the other half will receive Standard of Care treatment

DETAILED DESCRIPTION:
One hundred and thirty-eight (138) subjects with chronic Diabetic Foot Ulcers ranging in size from 1cm2 to 25cm2 will be randomized 1:1 to either SynPath™ or Standard of Care after the completion of a 14 day screening/run-in period. Following the of run-in period the subjects with a 'hard to heal' or chronic, (>4 weeks) nonresponsive Wagner Grade 1 or 2 diabetic foot ulcer will be randomized to receive either SynPath™ or SOC treatment. Both treatment groups will require subjects to use off-loading device.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. A signed and dated informed consent form has been obtained from the subject
3. Confirmed Type 1 or 2 diabetes with a hemoglobin HbA1c ≤12% within 90 days of informed consent
4. Current reference ulcer has been in existence for longer than four (4) weeks with confirmed failure of a prior treatment to heal the ulcer, prior to signing informed consent for trial participation. Verbal statement from prior treating clinician or patient can be used as confirmation of treatment failure.
5. Reference ulcer has been diagnosed as either a partial or full thickness diabetic foot ulcer without tunneling, undermining, sinus tracts or /exposed bone, with a scale rating of a Wagner Grade 1 or Wagner Grade 2 extended to ligament, tendon, and joint capsule with no bone exposure
6. Ulcer is either located on the foot or ankle with at least 50% of ulcer below medial aspect of the malleolus
7. Ulcer size (area) ≥1cm² and ≤25cm² post-debridement at both screening visit 1 and at baseline/randomization visit 3
8. There is a minimum 1cm margin between the qualifying reference study ulcer and any other ulcers on the specified foot, post debridement
9. Subject has adequate vascular perfusion of the affected limb, as defined by at least one of the following:

   1. Ankle-brachial Index (ABI) ≥ 0.65 or ≤1.2
   2. Toe pressure (plethysmography) >50mmHg
   3. TcPO2 >40mmHg
   4. Or as an alternative, the arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle or a TBI (Toe Brachial Index) of > 0.6 is acceptable.
10. Subject or responsible caregiver is willing and able to adhere to schedule of required applicable dressing changes as well as off-loading for the location of the reference ulcer
11. Subject is able and willing to comply with study procedures
12. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence) during the course of the study and undergo pregnancy tests.
13. A two-(2) week run-in period will Standard of Care treatment plus required offloading precede randomization in the trial to document the indolent nature of the subject's selected selected. The subject may be randomized if the reference ulcer has not reduced in area >30% from screening visit 1 to baseline/randomization visit 3.

Exclusion Criteria:

1. Subject was previously randomized and treated under this clinical study protocol
2. Subject has suspected or confirmed signs/symptoms of gangrene or wound infection as evidenced by redness, pain, and purulent drainage on any part of the index limb as confirmed by X-ray or biopsy
3. Subject has a history of hypersensitivity to polyurethane, as determined by prior medical history
4. Subject has participated in another clinical trial involving a device or a systemically administered investigational study drug/treatment within 30 days of randomization
5. Subject has received, or is scheduled to receive a medication or treatment which is known to interfere with or affect the rate or quality of wound healing within 30 days of signing the informed consent form
6. Subject has a history of bone cancer or metastatic disease on the index limb, radiation therapy to the foot, or has had chemotherapy within twelve (12) months prior to signing informed consent form for trial participation
7. Reference ulcer, in the clinical opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer
8. Subject has a condition that would interfere with their ability to adhere with the treatment regimen or has a known history of poor adherence with medical treatment
9. In the opinion of the Investigator, the subject has a history of or is currently diagnosed with any illnesses or conditions, other than diabetes, that could interfere with wound healing such as auto-immune disorders, end-stage renal disease, severe malnutrition, liver disease or connective tissue disorders
10. In the clinical opinion of the Investigator, the subject has an active or unstable Charcot foot
11. Subject has ulcers secondary to a disease other than diabetes (e.g., vasculitis, neoplasms, or hematological disorders)
12. In the clinical opinion of the Investigator, the subject has excessive lymphoedema that could interfere with off-loading and/or wound healing
13. Subject with an active infection at the reference ulcer
14. Subject has a non-healed surgical site from a prior amputation located in the index limb that has been open for less than 30 days
15. Subject has been treated with wound dressings that include growth factors, engineered tissues or skin substitutes within 30 days of randomization or is scheduled to receive treatment during the study
16. Subject has been treated with hyperbaric oxygen or topical oxygen therapy within five (5) days of the Screening Visit or is scheduled to receive hyperbaric oxygen treatment or topical oxygen therapy during the study
17. Subject has been treated with Negative Pressure Wound Therapy (NPWT) within 72 hours of the Screening Visit
18. Subject receiving dialysis treatment: hemodialysis or peritoneal dialysis
19. Subject has received an organ transplant
20. Subjects with a history of more than two (2) weeks treatment with immunosuppressants including prednisone 10 mg daily or an equivalent dose of other oral steroids, or application of topical steroids to the ulcer surface within one (1) month prior to first Screening Visit, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study
21. Active osteomyelitis or bone infection of the index foot. A subject may be enrolled in study if the subject:

    1. is at least 8 weeks post osteomyelitis diagnosis
    2. has been treated appropriately
    3. has only intact joint capsule exposed with no bone exposure
22. Subjects presenting with an ulcer probing to bone (Wagner Grade 3)
23. Subject is currently pregnant or actively trying to conceive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Percentage of ulcer closed at 12 weeks | 12 weeks
  Complete wound closure was defined as 100% re-epithelialization of the ulcer surface without drainage or dressing requirements confirmed at 2 consecutive study visits 2 weeks apart

SECONDARY OUTCOMES:
Percentage of ulcers that achieved 50% or greater closure rate within 6 weeks | 6 weeks
  The percentage of ulcers that achieve 50% or greater closure
Comparison of closure rates for each treatment group | 12 weeks
  Comparison of rates of wound closure between Standard of Care and SynPath
Percent Wound Area Reduction(PWAR) over 12 weeks | 12 Weeks
  The Change in percentage wound reduction(PWVR) over 12 weeks for each treatment group
Cost of treatment in each treatment group | 12 weeks
  Calculation of cost of treatment including number of device applications for each treatment group
Change in reported Pain Levels between each treatment group | 12 weeks
  Change in subject reported pain levels using the 0-10 Numerical Pain Scale
The type and number of serious adverse events experienced | 12 weeks
  Comparison of the type and number of serious adverse events experience for each treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Zelen, DPM, FACFAC, Study Director — Profession Education and Research Institute, LLC
Locations (7):
- United States (7):
  - Center for Clinical Research, Castro Valley, California
  - Limb Preservation Platform, Inc, Fresno, California
  - ILD Research Center, Vista, California
  - Barry University Clinical Research, Tamarac, Florida
  - Lower Extremity Institute for Research and Therapy, LLC, Youngstown, Ohio
  - JPS Health Network, Fort Worth, Texas
  - Foot and Ankle Specialists of Mid-Atlantic, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No